CLINICAL TRIAL: NCT00336869
Title: Partnership Programs to Reduce Cardiovascular Disparities- Morehouse- Emory Partnership
Acronym: Meta-Health
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Morehouse School of Medicine (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Other Study IDs: IRB00024856; 1024-2004 (Other: Other)
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples metabolic testing

SUMMARY:
The theme of this Morehouse-Emory Partnership Program focuses on elucidating the etiologic basis of ethnic differences in obesity-related CVD and discovering new intervention strategies to ameliorate CV health in all communities. The proposed Program uses a multi-disciplinary strategy to systematically characterize ethnic differences in obesity-related CVD by drawing upon the fields of physiology, psychology, biochemistry, vascular biology, public health, nursing and clinical medicine.

DETAILED DESCRIPTION:
Emerging evidence indicates that there are ethnicity-specific differences in the profile of biochemical, metabolic and physiological perturbations associated with obesity. The implications of these ethnic differences remain to be further defined. Several epidemiologic studies have shown that vascular disease and its cardiovascular complications, carry significantly higher morbidity and mortality in African Americans compared with Caucasians.1-3 These observations may be partly explained by a higher prevalence of cardiovascular disease risk factors, such as essential hypertension, diabetes mellitus, and tobacco use among African Americans.4-6 However, the pathophysiological processes underlying this racial predisposition have not been fully elucidated.7 It is likely that the etiologic basis of ethnic disparities in cardiovascular disease is multi-factorial and involves dynamic gene-environment interactions in which variances in behavior and the social context are critical determinants.

The proposed Program recognizes the importance of incorporating both biological factors and social determinants in the analysis of cardiovascular disparities

ELIGIBILITY:
Inclusion Criteria:

Our methodological approach will involve a random digit-dialing cross-sectional survey of 4000 Metro Atlanta area AA and white residents (ages 30-65 years). This aim will focus on using well-validated survey instruments to examine self-reported perceptions of psychosocial stress, neighborhood segregation factors and health beliefs related to weight/weight control. These parameters will be assessed in relation to the differential prevalence of three major outcomes: (1) self-reported maladaptive cardiovascular behaviors that predispose to obesity-related CVD (ie high fat/sodium and low fruit/vegetables dietary intake and physical inactivity); (2) obesity; and (3) hypertension.

This study will address the following research questions: Are the observed racial differences in maladaptive health behaviors (diet/inactivity) and MetS components (obesity, hypertension) associated with: a) perceived psychosocial stress, and if so, does depression, neighborhood factors or health beliefs around weight and weight control modify this relationship?

-

Exclusion Criteria:

-

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African American and White residents age 30-65
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University; Gary Gibbons, MD, Principal Investigator — Morehouse School of Medicine
Locations (2):
- United States (2):
  - Morehouse CRC, Atlanta, Georgia
  - Emory GCRC, Atlanta, Georgia